CLINICAL TRIAL: NCT00516724
Title: A Phase I, Open-Label Study to Assess the Safety and Tolerability of KU-0059436 in Combination With Carboplatin, KU-0059436 in Combination With a Paclitaxel/Carboplatin T/C Doublet and KU-0059436 in Combination With Paclitaxel in the Treatment of Patients With Advanced Solid Tumours
Brief Title: Study to Assess the Safety and Tolerability of a PARP Inhibitor in Combination With Carboplatin and/or Paclitaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KU36-96; D0810C00004; 2007-000939-26 (EudraCT Number)
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Triple Negative Metastatic Breast Cancer; Advanced Ovarian Cancer; Carboplatin; Paclitaxel
Keywords: malignant solid tumours; Poly(ADP ribose) polymerases
MeSH Terms: interventions — olaparib; Carboplatin; Paclitaxel; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Carboplatin + KU-0059436
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor); Drug: Carboplatin
- 2. (Experimental): Paclitaxel + KU-0059436
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor); Drug: Paclitaxel
- 3. (Experimental): Paclitaxel, Carboplatin + KU-0059436
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor); Drug: Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib
  Arms: 1
Drug: Carboplatin — intravenous injection
  Other Names: CBDCA; Paraplatin®
  Arms: 1
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — Oral
  Other Names: Olaparib
  Arms: 2.
Drug: Paclitaxel — Intravenous injection
  Arms: 2.
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — Oral
  Other Names: Olaparib
  Arms: 3.
Drug: Paclitaxel + Carboplatin — Intravenous injection
  Arms: 3.

SUMMARY:
The purpose of this study is to identify a safe and tolerable dose of the drug KU-0059436 that can be given in combination with carboplatin and/or Paclitaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a histologically or cytologically diagnosed malignant solid tumour
* Adequate bone marrow, hepatic and renal function
* Performance status of no more than 2 ( ECOG scale).

Exclusion Criteria:

* Any chemotherapy, radiotherapy ( except palliative), endocrine or immunotherapy within 4 weeks prior to entry
* Major surgery with 4 weeks of entering the study and must have recovered from effects of the major surgery
* More than two previous courses of platinum-containing chemotherapy
* Heavily pre-treated patients(> 2 courses of previous chemotherapy and/or extensive irradiation leading to bone marrow deficiency) will be excluded from the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2007-06-22 (Actual); Primary Completion 2013-01-04 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of KU 0059436 in combination with Paclitaxel/Carboplatin | assessed at each visit

SECONDARY OUTCOMES:
To identify the dose limiting toxicity of the combination therapy | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Dr Johann de Bono, MD, Principal Investigator — Cancer Research UK, The Institute of Cancer Research, London, UK; Prof Jan HM Schellens, Principal Investigator — The Netherlands Cancer Institute, Amsterdam, The Netherlands
Locations (4):
- Research Site, Brussels, Belgium
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] van der Noll R, Jager A, Ang JE, Marchetti S, Mergui-Roelvink MWJ, Lolkema MP, de Jonge MJA, van der Biessen DA, Brunetto AT, Arkenau HT, Tchakov I, Beijnen JH, de Bono JS, Schellens JHM. Phase I study of continuous olaparib capsule dosing in combination with carboplatin and/or paclitaxel (Part 1). Invest New Drugs. 2020 Aug;38(4):1117-1128. doi: 10.1007/s10637-019-00856-7. Epub 2019 Oct 30. PMID 31667659
- [Derived] van der Noll R, Jager A, Ang JE, Marchetti S, Mergui-Roelvink MWJ, de Bono JS, Lolkema MP, de Jonge MJA, van der Biessen DA, Brunetto AT, Arkenau HT, Tchakov I, Beijnen JH, De Greve J, Schellens JHM. Phase I study of intermittent olaparib capsule or tablet dosing in combination with carboplatin and paclitaxel (part 2). Invest New Drugs. 2020 Aug;38(4):1096-1107. doi: 10.1007/s10637-019-00857-6. Epub 2019 Oct 21. PMID 31637669
- [Derived] Shamseddine AI, Farhat FS. Platinum-based compounds for the treatment of metastatic breast cancer. Chemotherapy. 2011;57(6):468-87. doi: 10.1159/000334093. Epub 2012 Jan 10. PMID 22248721
- See also: KU36-96_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2679&filename=CSR_Synopsis_D0810C00004(KU36-96).pdf
- See also: revised_CSP9 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=KU36-96&attachmentIdentifier=9f78dafb-adbe-406e-92e2-30b9ed9a532b&fileName=KU3696__RevisedCSP9_redacted_SECURE.pdf&versionIdentifier=
- See also: Study Results — https://www.astrazenecaclinicaltrials.com/study/KU36-96/